CLINICAL TRIAL: NCT04719104
Title: Can Transcutaneous Bilirubin (TcB) Measurements be Utilised to Assess Rebound Hyperbilirubinaemia Following Phototherapy in Neonates?
Brief Title: Transcutaneous Bilirubin Measurements in Neonates Post Phototherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GN20HP515
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Jaundice, Neonatal
Keywords: Jaundice; Neonate; Transcutaneous; Phototherapy; Bilirubin
MeSH Terms: conditions — Jaundice, Neonatal; Jaundice

STUDY DESIGN:
Intervention Model Description: The study population will include 200 newborns of 35 weeks' gestation or greater who are over 24 hours old. Each baby will be studied only once.
  In addition to the routine SBR (capillary blood sample to measure serum bilirubin (jaundice), a paired TcB measurement will be taken 10-14 hours after stopping phototherapy. Taking a TcB measurement will involve using a 'biliflash'. This is a non-invasive measurement that flashes a light against the baby's ear and can be done at the cotside. The test takes less than a minute and does not cause the baby discomfort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participating group of neonates (Experimental): Participating group: Neonates that have had both a serum bilirubin measurement and transcutaneous measurement post phototherapy. This is a single arm study as we are only targeting one group of individuals with the intervention (transcutaneous bilirubin measurement). However, we will compare the serum bilirubin measurement to the transcutaneous measurement from the same neonate to determine if there is a clinically significant difference between the two measurements.
  Interventions: Device: Transcutaneous Bilirubin Meter - 'Bilimeter'

INTERVENTIONS:
Device: Transcutaneous Bilirubin Meter - 'Bilimeter' — Taking a transcutaneous (TcB) measurement will involve using a 'biliflash'. This is a non-invasive measurement that involves flashing a light against the helix of the infant's ear and can be done at the cotside. This process takes approximately 1-2 minutes and does not cause the baby discomfort. The meter gives an immediate bilirubin level.

SUMMARY:
Can transcutaneous bilirubin (TcB) measurements be utilised to assess rebound hyperbilirubinaemia following phototherapy in neonates?

DETAILED DESCRIPTION:
Jaundice is common in the newborn and may result in the need for babies to be readmitted from home for phototherapy, with associated increased costs and significant family distress.

As well as prolonged hospital stay, neonates on phototherapy require multiple blood tests (SBR), generally acquired via heel prick testing. These cause the baby discomfort and samples may be insufficient or haemolyzed and require repeating. There is also a delay of one to two hours at best in results being received and actioned.

Jaundice measurements can also be obtained using non-invasive, cheap and reliable meters (TcB) that give almost immediate results. The meter takes one to two minutes to get a result and can be used at the cotside. TcB causes the baby no significant discomfort.

TcB meters are commonly used before phototherapy but are not routinely used during or after stopping phototherapy. Jaundice commonly worsens after stopping phototherapy due to release of bilirubin from tissues and so measuring a "rebound" SBR twelve hours after stopping phototherapy and before the baby can go home is routine practice.

TcB meters tend to underestimate SBR in the first eight hours after stopping phototherapy but there is some evidence that thereafter they may provide reliable results. If TcB measurements can be used as a reliable predictor for SBR twelve hours after phototherapy, this will reduce blood sampling and costs, causing less distress to the baby and their mother, with potential for earlier discharge home. The NICE guideline for neonatal jaundice suggests that new research is needed to evaluate the accuracy of different transcutaneous bilirubinometers in comparison to serum bilirubin levels in all babies.

ELIGIBILITY:
Inclusion Criteria:

* Well neonates
* 35+0 weeks gestation or greater, over 24 hours old
* Inpatients at Princess Royal Maternity (PRM), NHS Greater Glasgow and Clyde

Exclusion Criteria:

* Unwell neonates
* Less than 35+0 weeks' gestation
* Less than 24 hours old
* Mother unable or too distressed to give informed consent

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Utility of transcutaneous bilirubinometer (TcB) in assessing rebound jaundice | 6 months
  Can the TcB be safely and effectively used to assess rebound hyperbilirubinaemia after phototherapy in babies of 35 weeks' gestation or greater?